CLINICAL TRIAL: NCT01607021
Title: Pharmacogenomics Study on IL28B Genetic Variants for Prediction of Drug Response in Chinese Children With HCV Infection.
Brief Title: Pharmacogenomics Study on IL28B Genetic Variants in Chinese Children With Hepatitis C Virus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: beijing302-004
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; interleukin 28; Children
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chinese children with HCV RNA positive: A sample of 200 children with a recent confirmation of anti-HCV-antibody positive and HCV RNA positive. All the children were treated with antiviral therapy, and the course of treatment depend on HCV Viral genotyping(ie, genotype 1,2,3,4 subtypes).
  Primary Outcome Measures:
  Virologic response [ Time Frame: Weeks 2, 4, 6, 8, 10, and 12 ] Sustained virologic response (SVR, defined as plasma HCV RNA < lower limit of quantification [LLoQ] at 24 weeks after treatment cessation) following antiviral treatment.
  Secondary Outcome Measures: Safety and tolerability of therapy. [ Time Frame: Up to 48 weeks ] measured by frequency of laboratory abnormalities , reported adverse events and discontinuations due to adverse events

SUMMARY:
The aim of this study is to investigate the relationships between interleukin 28B genetic variants and the response to treatment of chronic hepatitis C in Chinese children.

DETAILED DESCRIPTION:
Hepatitis C affects thousands of children throughout the world. Most children acquire the virus through vertical transmission, although parenteral routes of acquisition are also common. Affected children are usually asymptomatic and histological findings are mild with a low risk of progression, about 5% develop significant liver disease in childhood.

The use of combination treatment with interferon-alpha and ribavirin were recommended in the treatment of chronic hepatitis C in children, SVR in children with genotype 1 ranged from 44% to 59%. SVR in children with genotype 2 and 3 was more than 90%. But both interferon and ribavirin have significant side effects which affect compliance, such as: repeated flu like symptoms, leukopenia and anemia, moderate weight loss, behavioural problems, thyroid dysfunction and transient deceleration of the growth rate. In addition, approximately 50% of children infected with genotype 1 do not respond to therapy.

Recent work has highlighted that single nucleotide polymorphisms (SNPs) around the IL28B gene have been identified as strong predictors of spontaneous and treatment-induced HCV clearance in adults, especially Rs 12979860 and Rs 8099917. A recent article in Hepatology also reported that interleukin (IL)-28B C/C genotype in the child was associated with spontaneous clearance of hepatitis C virus (HCV) genotype 1 infection. All this reports show that Genetic Variation in Interleukin-28B Locus is associated with the procession of CHC.

The aim of this study was to study the association between genetic variation in IL-28B and the development of CHC in Chinese children, such as: HCV viral load, serum alanine aminotransferase, histological change and the response to the treatment with interferon-alpha and ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1-18 years
* Patients with chronic HCV infection

Exclusion Criteria:

* HCV infected patients previously treated with antiviral drugs
* Co-infected Patients with HIV or Hepatitis B virus (HBsAg positive)
* hepatocellular carcinoma or other malignancies
* anticipated with difficulty of follow-up observation

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 200 children with chronic HCV infection who were seen at beijing 302 hospital(Beijing China)between april 2012 and december 2012.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: jin han, professor, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, Beijing Municipality, China